CLINICAL TRIAL: NCT04156945
Title: Interventions to Curb Hepatitis C Reinfections Among Men Who Have Sex With Men
Acronym: ICECREAM
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Public Health Service of Amsterdam (Other Government)
Collaborators: ZonMw: The Netherlands Organisation for Health Research and Development (Other); Amsterdam University Medical Centers (UMC), Location Academic Medical Center (AMC) (Other); The National Institute for STI and Aids Control in the Netherlands (Soa Aids Nederland) (Unknown); Julius Centre for Health Sciences and Primary Care, UMC Utrecht (Unknown); ANRS | Maladies infectieuses émergentes (Unknown)
Responsible Party: Principal Investigator, Prof. dr. Maria Prins, Prof. dr., Public Health Service of Amsterdam
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: NL68718.018.19
Record Dates: First submitted 2019-10-07; First posted 2019-11-08 (Actual); Last update posted 2024-08-02 (Actual); Status verified 2024-08

CONDITIONS: Hepatitis C Virus Infection
Keywords: Hepatitis C virus (HCV) reinfection; Men who have sex with men (MSM)
MeSH Terms: conditions — Hepatitis C; Reinfection; Homosexuality

STUDY DESIGN:
Intervention Model Description: A 3-arm multicenter randomized trial. The trial will start with a 6 month run-in period (standard care) to determine at-risk behaviour under no intervention.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Intervention I: behavioural intervention (Experimental): Participants will receive the behavioural Intervention in addition to standard of care.
  Interventions: Behavioral: Behavioural intervention
- Intervention II: home-based testing intervention (Experimental): Participants will receive the home-based testing intervention in addition to standard of care.
  Interventions: Diagnostic Test: HCV RNA home-based test
- Intervention III: combined intervention (Experimental): Participants will receive the behavioural intervention and the home-based testing intervention in addition to standard of care.
  Interventions: Behavioral: Behavioural intervention; Diagnostic Test: HCV RNA home-based test

INTERVENTIONS:
Behavioral: Behavioural intervention — An online tailored behavioural intervention. The intervention will be developed as part of the project and will be based on the principles of the Information-Motivation-Behavioural Skills (IBM) model for behavioural change. It will consist of four interactive text-based modules, and demonstration and modelling videos addressing information, motivation, and behavioural skills. The intervention will be offered on a website and able to be used on PCs as well as any mobile device. It will be provided to the participants after randomization at month 6 and available for a total period of 18 months.
  Arms: Intervention I: behavioural intervention; Intervention III: combined intervention
Diagnostic Test: HCV RNA home-based test — An additional patient-initiated home-based HCV testing service. The service offers a maximum of 4 free-of-charge HCV-RNA tests, which involves HCV testing using self-sampled dried blood spots (DBS). The DBS obtained from a finger stick will be used for HCV-RNA testing in the laboratory. DBS test kits, along with instructions and package materials for returning the test kits with the self-collected DBS sample will be provided to the participants after randomization at month 6 and available for use for a total period of 18 months.
  Arms: Intervention II: home-based testing intervention; Intervention III: combined intervention

SUMMARY:
Men who have sex with men (MSM) who cured from hepatitis C virus (HCV) infection are at substantial risk of HCV reinfection. In this study, the investigators aim to evaluate the effectiveness of an online behavioural intervention, a home-based testing intervention and a combination of both on risk behaviour, and ultimately preventing HCV reinfection and onward spread of HCV.

DETAILED DESCRIPTION:
Rationale: As highly effective therapy against hepatitis C virus (HCV) infection is available with rapid uptake, there is newfound optimism for HCV elimination. Nevertheless, HCV reinfections cause great concern in at risk populations, including men who have sex with men (MSM). In the Netherlands, MSM account for the majority of new HCV (re)infections. Although HCV treatment uptake is high in this group, modelling data indicate HCV elimination would not be feasible without a reduction in risk behaviour. This finding highlights the urgent need for effective interventions aimed at reducing risk behaviour and preventing reinfections in MSM.

Objective: To evaluate interventions aimed at reducing risk behaviour, and ultimately preventing HCV reinfections and onward spread of HCV.

Study design: Using a 3-arm randomised trial comparing run-in and intervention periods, we will evaluate the effect of two interventions and its combination on risk behaviour in MSM previously infected with HCV.

Study population: MSM aged 18 years or older with a history of a successfully treated or spontaneously cleared HCV infection.

Interventions: Intervention I is a targeted, online behavioural intervention developed as part of the project. Intervention II aims to increase the frequency of testing by offering an additional patient-initiated, home-based HCV RNA testing service with the use of self-sampled dried blot spots. Intervention III is a combination of intervention I and II.

Study parameters/endpoints: From run-in and post-randomization questionnaires, we will evaluate the proportion at risk of HCV infection (as determined by the HCV-MOSAIC score) as the primary outcome. The HCV-MOSAIC risk score is calculated by summing up the beta coefficients specific to six self-reported risk factors when present: receptive condomless anal sex (beta 1.1), sharing sex toys (beta 1.2), unprotected fisting (beta 0.9), injecting drug use (beta 1.4), sharing straws during nasally-administered drug use (beta 1.0), and ulcerative sexually transmitted infection (beta 1.4). Secondary outcomes include incidence of HCV reinfection, changes in the individual risk behaviour items and changes in sexual wellbeing.

ELIGIBILITY:
Inclusion Criteria:

* Informed consent documented by signature.
* Male individual aged 18 years or older.
* History of a cured or spontaneously cleared HCV infection (positive HCV RNA test in the past and/or positive anti-HCV IgG).
* Self-reported MSM who are either (i) HIV-positive seeking care at an HIV treatment center or (ii) HIV-negative and seeking care at an STI/PrEP/sexual health center.
* Sufficient understanding of Dutch or English.
* Have internet access and an e-mail address.

Exclusion Criteria:

* Acute or chronic HCV infection at time of enrolment.
* Under HCV treatment at time of enrolment.
* Unlikely, in the opinion of the clinician, to comply with the study procedures.
* Currently participating in an intervention study that offers extra HCV testing and/or a behavioural intervention targeting risk behaviour.
* Investigators or otherwise dependent persons.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Men who have sex with men (MSM)
Enrollment: 258 (Actual)
Dates: Start 2021-09-14 (Actual); Primary Completion 2026-02 (Estimated); Study Completion 2026-02 (Estimated)

PRIMARY OUTCOMES:
Change in the proportion at risk for HCV infection (as determined by a HCV-MOSAIC risk ≥ 2.0). | Run-in period (0-6 months) versus intervention period (6-24 months)
  From run-in and post-randomization questionnaires, we will evaluate the proportion at risk of HCV infection (as determined by a HCV-MOSAIC score ≥ 2.0) during the run-in versus intervention periods. The HCV-MOSAIC risk score has been previously validated for acute HCV-infection and is calculated by summing up the beta-coefficients specific to six self-reported risk factors when present in the past 6 months: (i) receptive condomless anal sex (beta 1.1), (ii) sharing sex toys (beta 1.2), (iii) unprotected fisting (beta 0.9), (iv) injecting drug use (beta 1.4), (v) sharing snoring equipment during nasally-administered drug use (beta 1.0), and (vi) ulcerative sexually transmitted infection (beta 1.4).

SECONDARY OUTCOMES:
Incidence rate of HCV reinfection. | Self-reported: month 0, month 6, month 12, month 18, month 24. Laboratory data: during total follow-up period of 2 years.
  Number of cases of HCV reinfection divided by total person-years of follow-up at risk for reinfection, self-reported and laboratory data.
Incidence rate of any STI. | Month 0, month 6, month 12, month 18, month 24
  Number of cases of chlamydia, gonorrhoea, lymphogranuloma venereum (LGV), genital herpes and/or syphilis divided by total person-years, self-reported.
Change in the number of sex partners. | Month 0, month 6, month 12, month 18, month 24
Change in the number of condomless anal sex acts with casual partners. | Month 0, month 6, month 12, month 18, month 24
Change in the proportion of individuals reporting receptive condomless anal sex. | Month 0, month 6, month 12, month 18, month 24
Change in the proportion of individuals sharing sex toys. | Month 0, month 6, month 12, month 18, month 24
Change in the proportion of individuals reporting unprotected fisting. | Month 0, month 6, month 12, month 18, month 24
Change in the proportion of individuals reporting injection drug use. | Month 0, month 6, month 12, month 18, month 24
Change in the proportion of individuals sharing snoring equipment during nasally-administered drug use. | Month 0, month 6, month 12, month 18, month 24
Change in the proportion of individuals reporting ulcerative sexually transmitted infection*. | Month 0, month 6, month 12, month 18, month 24
  *syphilis, genital herpes or lymphogranuloma venereum infection
Proportion of individuals with change in any of the items of the HCV-MOSAIC risk score. | Month 0, month 6, month 12, month 18, month 24
Change in the frequency of recreational drug use before and during sex. | Month 0, month 6, month 12, month 18, month 24
Change in the frequency of individuals engaging in group sex activities, including changes in number of events and maximum number of sex partners during an event. | Month 0, month 6, month 12, month 18, month 24
Change in the proportion of individuals sharing lubricants. | Month 0, month 6, month 12, month 18, month 24
Change in the proportion of individuals sharing anal douches. | Month 0, month 6, month 12, month 18, month 24
Change in the proportion of individuals disinfecting sex toys, skin and/or sex location. | Month 0, month 6, month 12, month 18, month 24
Change in sexual wellbeing score. | Month 0, month 6, month 12, month 18, month 24

OTHER OUTCOMES:
Characteristics of the study population (e.g. age, etnicity, hiv-status) | Month 0
The proportion of individuals reporting change in the risk behaviour identified in the goal setting module of the behavioural intervention. | During the intervention period, month 6 until month 24
Website statistics (e.g., frequency of use, time spent on the behavioural intervention and the proportion of individuals completing all modules of the intervention). | During the intervention period, month 6 until month 24
Type of goals set in the behavioural intervention. | During the intervention period, month 6 until month 24
Usability and acceptability of the behavioural intervention. | During the intervention period, month 6 until month 24
The proportion of free HCV tests used (the total number of free HCV tests used divided by the total number of distributed tests). | During the intervention period, month 6 until month 24
The proportion of HCV positive test results (the total number of HCV positive test results divided by the total number of free tests used). | During the intervention period, month 6 until month 24
Usability and acceptability of the testing intervention. | During the intervention period, month 6 until month 24
The number of (home-based) tests obtained and used from other sources. | Month 0, month 6, month 12, month 18, month 24

CONTACTS AND LOCATIONS:
Overall Officials: Maria Prins, Prof. dr., Principal Investigator — Public Health Service of Amsterdam (GGD Amsterdam)
Locations (15):
- France (5):
  - Le Centre 190, Paris
  - Maison Chemin Vert, Paris
  - Service de maladies infectieuses et tropicales, Hôpital La Pitié-Salpêtrière, Paris
  - Service de maladies infectieuses et tropicales, Hôpital Saint-Antoine, Paris
  - Service de maladies infectieuses et tropicales, Hôpital Tenon, Paris
- Netherlands (10):
  - Public Health Service of Amsterdam (GGD Amsterdam), Amsterdam, North Holland
  - Onze Lieve Vrouwe Gasthuis locatie West, Amsterdam, North Holland
  - DC Klinieken Lairesse, Amsterdam, North Holland
  - Medisch Centrum Jan van Goyen, Amsterdam, North Holland
  - Vrije Universiteit Medisch Centrum, Amsterdam, North Holland
  - Onze Lieve Vrouwe Gasthuis locatie Oost, Amsterdam, North Holland
  - Amsterdam UMC - locatie AMC, Amsterdam, North Holland
  - Maasstad Ziekenhuis, Rotterdam, South Holland
  - Haaglanden Medisch Centrum, The Hague, South Holland
  - Universitair Medisch Centrum Utrecht, Utrecht

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Newsum AM, Stolte IG, van der Meer JT, Schinkel J, van der Valk M, Vanhommerig JW, Buve A, Danta M, Hogewoning A, Prins M; MOSAIC collaborators. Development and validation of the HCV-MOSAIC risk score to assist testing for acute hepatitis C virus (HCV) infection in HIV-infected men who have sex with men (MSM). Euro Surveill. 2017 May 25;22(21):30540. doi: 10.2807/1560-7917.ES.2017.22.21.30540. PMID 28597832
- [Background] Lambers FA, Prins M, Thomas X, Molenkamp R, Kwa D, Brinkman K, van der Meer JT, Schinkel J; MOSAIC (MSM Observational Study of Acute Infection with hepatitis C) study group. Alarming incidence of hepatitis C virus re-infection after treatment of sexually acquired acute hepatitis C virus infection in HIV-infected MSM. AIDS. 2011 Nov 13;25(17):F21-7. doi: 10.1097/QAD.0b013e32834bac44. PMID 21857492
- [Background] Lambers F, van der Veldt W, Prins M, Davidovich U; MOSAIC study. Changing the odds: motives for and barriers to reducing HCV-related sexual risk behaviour among HIV-infected MSM previously infected with HCV. BMC Infect Dis. 2018 Dec 18;18(1):678. doi: 10.1186/s12879-018-3571-1. PMID 30563503
- [Derived] Hage K, Boyd A, Davidovich U, Zantkuijl P, Hoornenborg E, Matser A, Generaal E, Schinkel J, Todesco E, van der Valk M, Rougier H, Lacombe K, Prins M; ICECREAM study group. Evaluating interventions to reduce behaviour associated with HCV reinfection in men who have sex with men: study protocol for a non-blinded, phase 2, randomised trial. Trials. 2023 Mar 15;24(1):193. doi: 10.1186/s13063-023-07161-y. PMID 36922871

DOCUMENTS (2):
  • Study Protocol (2022-03-17): https://cdn.clinicaltrials.gov/large-docs/45/NCT04156945/Prot_001.pdf
  • Statistical Analysis Plan (2023-06-01): https://cdn.clinicaltrials.gov/large-docs/45/NCT04156945/SAP_002.pdf